CLINICAL TRIAL: NCT02007577
Title: Beneficial Effect of Salicylates: Insulin Action, Secretion or Clearance?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Gerald M Reaven, Professor Emeritus, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 19254
Record Dates: First submitted 2013-03-05; First posted 2013-12-11 (Estimated); Results first posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Pre Diabetes; Insulin Resistant
Keywords: insulin resistant
MeSH Terms: conditions — Glucose Intolerance | interventions — salicylsalicylic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- salsalate 3500mg in 2 divided doses a day (Active Comparator): Participants will take 3, 500 mg tablets with breakfast and 4, 500 mg tablets with dinner
  Interventions: Drug: salsalate
- placebo (Placebo Comparator): Participants will take 3 placebo tablets with breakfast and 4 placebo tablets with dinner
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: salsalate — Participants will take 3, 500 mg tablets with breakfast and 4, 500 mg tablets with dinner
  Arms: salsalate 3500mg in 2 divided doses a day
Drug: Placebo — Participants will take 3 tablets with breakfast and 4 tablets with dinner
  Arms: placebo

SUMMARY:
The possibility that obesity-associated inflammatory changes may play a role in the pathogenesis of type 2 diabetes (2DM) has led to increased interest in the possibility that salicylates might represent a useful treatment to improve glucose tolerance. Several studies, performed in patients with 2DM, as well as in nondiabetic, obese individuals, have demonstrated that salicylates have beneficial effects on glucose and insulin metabolism, but have not led to a coherent view as to the mechanism(s) involved.

In this research proposal we will use specific methods to quantify insulin mediated glucose uptake (IMGU), glucose-stimulated insulin secretion rate (GS-ISR), and insulin clearance (I-Cl) in overweight/obese, nondiabetic, insulin resistant individuals. We will use the insulin suppression test (IST) to quantify IMGU in nondiabetic, overweight/obese volunteers to identify those individuals who are sufficiently insulin resistant to be enrolled in this study. We will then use the graded glucose infusion technique in these insulin resistant subjects to generate specific measures of both GS-IS and I-Cl. Following these baseline measurements, salsalate or placebo will be administered for one month to the participants, after which time the IST and the graded glucose infusion will be repeated to quantify and compare the changes in IMGU, GS-ISR, and I-Cl that have resulted from salsalate versus placebo. These results will provide for the first time quantitative data of the effect of salicylates on IMGU, GS-ISR, and I-Cl in overweight/obese, insulin resistant, nondiabetic individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers,
* BMI 25-35kg/m2,
* Without severe anemia, kidney, liver disease or any current GI ulcers or bleeding
* Or on any medication contraindicated with salsalate

Exclusion Criteria:

* Recent history of GI bleed or ulcers,
* CVD or on anticoagulants
* Severe kidney or liver disease
* Allergies to aspirin
* Taking aspirin or anti inflammatory medication on a regular basis and cannot be taken off for the duration of the study

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2010-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald M Reaven, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim SH, Liu A, Ariel D, Abbasi F, Lamendola C, Grove K, Tomasso V, Ochoa H, Reaven G. Effect of salsalate on insulin action, secretion, and clearance in nondiabetic, insulin-resistant individuals: a randomized, placebo-controlled study. Diabetes Care. 2014 Jul;37(7):1944-50. doi: 10.2337/dc13-2977. PMID 24963111

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Salsalate 3500mg in 2 Divided Doses a Day | Placebo
Started | 27 | 14
Completed | 26 | 13
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Salsalate 3500mg in 2 Divided Doses a Day | Placebo | Total
Number analyzed (Participants) | 26 | 13 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10) | 54 (10) | 54 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 14 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: Quantification of Insulin Action With the Insulin Suppression Test (IST)
Description: Compare changes in insulin sensitivity as assesses by the IST before and after treatment between salsalate and placebo group
Time Frame: after treatment for one month
Measure: Median (95% Confidence Interval); unit: mmol/L
Arm/Group | Salsalate 3500mg in 2 Divided Doses a Day | Placebo
Number analyzed (Participants) | 26 | 13
mmol/L | -3 [-10 to 5] | 2 [-9 to 12]

2. Secondary Outcome: Quantification of Insulin Clearance With the Graded Glucose Infusion Test (GGIT)
Description: compare changes in insulin clearance as assessed by the GGIT before and after treatment with salsalate to placebo
Time Frame: one month on treatment
Measure: Median (95% Confidence Interval); unit: pmol/min x 4h
Arm/Group | Salsalate 3500mg in 2 Divided Doses a Day | Placebo
Number analyzed (Participants) | 26 | 13
pmol/min x 4h | -6 [-12 to 0] | 0 [-9 to 9]

ADVERSE EVENTS:
Arm/Group | Salsalate 3500mg in 2 Divided Doses a Day | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/14
Other Adverse Events (participants affected / at risk) | 1/27 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salsalate 3500mg in 2 Divided Doses a Day (N=27) | Placebo (N=14)
3 years (Gastrointestinal disorders) | 1 (1) | 0 (0) — heartburn
tinnitus (Ear and labyrinth disorders) | 1 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes